CLINICAL TRIAL: NCT01420978
Title: High Volume Cerebrospinal Fluid Diversion in the Management of Aneurysmal Subarachnoid Hemorrhage: A Pilot Study
Brief Title: Cerebrospinal Fluid (CSF) Drainage Study
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Responsible Party: Principal Investigator, Giuseppe Lanzino, MD, Mayo Clinic
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 11-002713
Record Dates: First submitted 2011-08-15; First posted 2011-08-22 (Estimated); Last update posted 2013-05-14 (Estimated); Status verified 2013-05

CONDITIONS: Aneurysmal Subarachnoid Hemorrhage
MeSH Terms: conditions — Subarachnoid Hemorrhage

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- High volume CSF diversion (Experimental): The EVD will be set to an initial level of 5 mmHg. The drain will remain in place at a level of ≤ 5 mmHg until at least day 10 after SAH before a weaning trial is attempted.
  Interventions: Procedure: CSF Diversion
- Conventional CSF diversion (Active Comparator): The EVD will be set to a level of 15 mmHg for as long as needed for the treatment of hydrocephalus, and subsequently weaned at the discretion of the treating physician. Lowering the level of the EVD can be considered by the treating physician if sustained intracranial hypertension occurs
  Interventions: Procedure: CSF Diversion

INTERVENTIONS:
Procedure: CSF Diversion — CSF drainage

SUMMARY:
When patients suffer a subarachnoid hemorrhage (bleeding around the brain), they often develop hydrocephalus. This is an enlargement of the fluid-filled spaces (ventricles) in the brain. Standard-of-care treatment includes placing an external ventricular drain (EVD) to drain off fluid. Eventually the EVD is weaned with the goal of removing it. Occasionally a patient does not tolerate this and a permanent surgery needs to be done to internalize a shunt.

Though this is done commonly and routinely throughout the world, there are no good studies to address how to optimally set the EVD level and how fast to wean it. Most set the EVD to a level of around 15 mmHg. The investigators hypothesize that setting the EVD lower (which will allow higher volume Cerebrospinal Fluid (CSF) drainage through the EVD) will improve perfusion at the level of the microcirculation in the brain, and result in improved neurologic outcomes.

ELIGIBILITY:
Inclusion Criteria

* Age ≥ 18 years
* Diagnosis of acute subarachnoid hemorrhage (SAH), confirmed with noncontrast head CT
* SAH is suspected to be aneurysmal in source
* Clinical management requires placement of EVD within 2 days of suspected time of hemorrhage

Exclusion Criteria

* Age < 18 years
* SAH of traumatic or non-aneurysmal etiology
* Patients treated with lumbar drains
* EVD placement ≥ 3 days after suspected time of hemorrhage
* Known contraindication to induction of relative intracranial hypotension (e.g. acute subdural hematoma)
* Pre-morbid mRS ≥ 3
* EVD that is suboptimally placed by CT obtained after EVD placement (i.e. EVD not in the ventricular system)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2011-08; Primary Completion 2013-02 (Actual); Study Completion 2013-02 (Actual)

PRIMARY OUTCOMES:
Modified Rankin Scale | 90-days
  The primary outcome is clinical outcome at 90 days. A favorable outcome is defined as a score of 1 or 2 on the modified Rankin Score (mRS) and poor outcome defined as a mRS of 3-6. This assessment will be made by a clinician who was blinded to the patient's CSF diversion treatment arm.

SECONDARY OUTCOMES:
Infarction | 90-days
  Presence of radiologic infarction
Vasospasm | 90-days
  Evidence of vasospams based upon TCD and/or angiography
Shunt placement | 90-days
  Rate of shunt placement
Ventriculitis | 90-days
  Rate of ventriculitis
Modified Rankin Scale | Hospital discharge (average 3 weeks)
  Modified rankin Scale upon discharge from the hospital
MMSE | 90-days
  Cognitive status evaluated using the MMSE
Length of ICU stay | Average 3 weeks
  Evalute the average length of ICU stay for this patient population.

CONTACTS AND LOCATIONS:
Overall Officials: Giuseppe Lanzino, MD, Principal Investigator — Mayo Clinic
Locations (2):
- United States (2):
  - Mayo Clinic in Florida, Jacksonville, Florida
  - Mayo Clinic in Rochester, Rochester, Minnesota